CLINICAL TRIAL: NCT07076472
Title: MC240704 Phase 1B Dose Escalation And Expansion Study of Sonodynamic Therapy With SONALA-001 in Combination With Exablate 4000 Type 2.0 MR-Guided Focused Ultrasound (MRgFUS) in Patients With Progressive or Recurrent Glioblastoma Multiforme (rGBM)
Brief Title: Sonodynamic Therapy With SONALA-001 and Magnetic Resonance Guided Focused Ultrasound for the Treatment of Progressive or Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240704; NCI-2025-04501 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-013192 (Other: Mayo Clinic Institutional Review Board); MC240704 (Other: Mayo Clinic); R44CA275508 (NIH)
Record Dates: First submitted 2025-07-15; First posted 2025-07-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Progressive Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SONALA-001, MRgFUS) (Experimental): Patients receive SONALA-001 IV over 15 minutes and undergo transcranial MRgFUS 3-8 hours after infusion on day 1 of each cycle. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a CT of the brain prior to treatment and blood sample collection and MRI throughout the study.
  Interventions: Drug: Aminolevulinic Acid Intravenous Formulation SONALA-001; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Magnetic Resonance Imaging; Procedure: MRI-Guided Focused Ultrasound Ablation

INTERVENTIONS:
Drug: Aminolevulinic Acid Intravenous Formulation SONALA-001 — Given IV
  Other Names: ALA Intravenous Formulation SONALA-001; SONALA 001; SONALA-001; SONALA001
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: MRI-Guided Focused Ultrasound Ablation — Undergo transcranial MRgFUS
  Other Names: Magnetic Resonance Imaging-guided High-Intensity Focused Ultrasound; Magnetic Resonance-guided Focused Ultrasound; MR-HIFU; MRgFUS; MRI Guided Focused Ultrasound Surgery; MRI-HIFU

SUMMARY:
This phase Ib trial tests the safety, best dose, and effectiveness of SONALA-001 in combination with magnetic resonance imaging-guided focused ultrasound (MRgFUS), also called sonodynamic therapy, in treating patients with glioblastoma that is growing, spreading, or getting worse (progressive) or that has come back after a period of improvement (recurrent). Sonodynamic therapy is a non-invasive combination therapy that uses low-intensity ultrasound, such as MRgFUS, to activate a drug, such as SONALA-001, to kill tumor cells. SONALA-001 binds to the tumor and may help the sonodynamic therapy target the tumor. MRgFUS is an image-guided, non-invasive technique that uses high energy ultrasound from the Exablate 4000 Type 2.0 device to kill tumors without damaging surrounding healthy tissue. Giving sonodynamic therapy using SONALA-001 with MRgFUS may be safe, tolerable, and/or effective in treating patients with progressive or recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize the safety, dose limiting toxicities (DLTs), maximum tolerated dose (MTD), maximum administered dose (MAD) and recommended phase 2 dose (RP2D) for future study after treatment with aminolevulinic acid intravenous formulation SONALA-001 (SONALA-001) in combination with MRgFUS in subjects with progressive or recurrent glioblastoma (rGBM).

SECONDARY OBJECTIVES:

I. To evaluate the preliminary antitumor activity as assessed by objective response rate (ORR; proportion of patients with complete or partial response) per Response Assessment in Neuro-Oncology (RANO) 2.0 guidelines.

II. To evaluate preliminary signals of activity as measured by clinical benefit rate (CBR) (proportion of patients with complete response, partial response or stable disease), progression-free survival (PFS), PFS rate at 6 months, and overall survival (OS).

OUTLINE:

Patients receive SONALA-001 intravenously (IV) over 15 minutes and undergo transcranial MRgFUS 3-8 hours after infusion on day 1 of each cycle. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a computed tomography (CT) of the brain prior to treatment and blood sample collection and magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 30 days, and then every 3 to 6 months for up to 3 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of recurrent or progressive glioblastoma (as defined in 2021 World Health Organization [WHO] Classification of Tumors of the Central Nervous System; Louis, Perry, et al. 2021) for which resection is not indicated as assessed by the study physician
* Radiographic evidence of disease which may be measurable or non-measurable
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Previous treatment with radiotherapy (RT)
* Have a life expectancy of ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 15 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 15 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (≤ 5 x ULN for patients with liver involvement) (obtained ≤ 15 days prior to registration)
* Albumin ≥ 3 g/dL (obtained ≤ 15 days prior to registration)
* Potassium ≥ lower limit of normal (LLN) (obtained ≤ 15 days prior to registration)
* Serum total calcium ≥ LLN (obtained ≤ 15 days prior to registration)
* Creatinine ≤ 1.5 x ULN OR calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault formula (obtained ≤ 15 days prior to registration)
* Negative pregnancy test done ≤ 8 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Willing to participate in the neuro-oncology biorepository [Institutional Review Board (IRB) 12-003458, principal investigator (PI): Jann Sarkaria, MD, PhD] for collecting and archiving biospecimens samples on neuro-oncology patients
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential (and persons able to father a child) who are unwilling to employ adequate contraception
* Recurrence ≤ 4 weeks after the completion of RT, defined from the imaging assessment immediately after completion of RT
* Three or more prior systemic treatments for recurrent or progressing disease
* Diagnosis of porphyria, or hypersensitivity to porphyrins
* Failure to recover to grade 1 or baseline from any adverse events (AEs) (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0) related to prior anticancer therapy

  * EXCEPTIONS: Alopecia, lymphopenia, peripheral neuropathy, and ototoxicity ≤ grade 3)
* Known history of the following conditions:

  * Allergy to gadolinium contrast agents
  * Patients known to be HIV positive and currently receiving antiretroviral therapy

    * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Inability to undergo MRI scans
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Patients with platelet count < 100
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  Defined per the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 as AEs considered to be at least possibly related to study treatment. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns (by dose level and overall).
Incidence of grade 3 or higher non-hematologic AEs | Up to 30 days after last dose of study treatment
  Defined per the CTCAE v5 as AEs considered to be at least possibly related to study treatment. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns (by dose level and overall).
Incidence of grade 4 or higher AE | Up to 30 days after last dose of study treatment
  Defined per the CTCAE v5 as AEs considered to be at least possibly related to study treatment. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns (by dose level and overall).
Dose-limiting event (DLE) | During first 6 weeks of therapy [first cycle of treatment (cycle length = 42 days)]
  AEs will be evaluated using CTCAE v5. The target DLE rate is < 33%.
Maximum tolerated dose (MTD) | Up to 6 weeks
  Will be defined as the highest safety-tolerated dose level where at most one patient out of six experiences a DLE.
Recommended phase 2 dose | Up to 6 weeks
  Will be determined based on a synthesis of safety, tolerability, clinical impact, patient response, and preliminary efficacy data from the initial dose and energy escalation stage.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 3 years
  Assessed by the proportion of patients with complete or partial response.
Clinical benefit rate | Up to 3 years
  Assessed by the proportion of patients with complete response, partial response or stable disease.
Progression-free survival (PFS) | Up to 3 years
  Defined as the time from registration to the earliest date of documentation of disease progression, relapse, or death due to any cause.
PFS at 6 months (PFS6) | At 6 months
  The PFS6 rate will be estimated as the number of patients who are progression-free and alive at 6 months.
Overall survival (OS) | Up to 3 years
  Defined as the time from registration to death due to any cause.
Time to response | Up to 3 years
  Defined as the time from registration to the first incidence of a response, estimated in patients who have achieved a response (PR or CR).
Duration of response | Up to 3 years
  Defined as the time from response to progression or death, whichever occurs first estimated among patients who have achieved objective response (PR or CR).
Duration of clinical benefit | Up to 3 years
  Defined as the time from response to progression or death, whichever occurs first, estimated among patients who achieved clinical benefit (stable disease, PR, or CR).

CONTACTS AND LOCATIONS:
Overall Officials: Terence C. Burns, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials